CLINICAL TRIAL: NCT06378177
Title: A Phase 2 Study of LVGN6051 Combined With Toripalimab and Paclitaxel for Recurrent/Metastatic HNSCC Rapidly Progressed From Previous Platinum-containing Curative Treatment or Contraindicated for Platinum-containing Treatment
Brief Title: A Study of LVGN6051 Combination Therapy in Patient With Head and Neck Squamous Cell Carcinoma (HNSCC)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Lyvgen Biopharma Holdings Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LVGN6051-0402-HNSCC
Record Dates: First submitted 2024-04-12; First posted 2024-04-22 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-04

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — toripalimab; Paclitaxel

STUDY DESIGN:
Intervention Model Description: This is a multicenter, open-labeled, single-arm Phase 2 clinical study.This study comprises two parts. Part 1 (Safety Run-in Phase) is designed to confirm the dose of combination therapy in Part 2.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LVGN6051combined with toripalimab and paclitaxel (Experimental): LVGN6051 in combination with toripalimab and paclitaxel
  Interventions: Biological: LVGN6051 Monoclonal Antibody Injection; Biological: toripalimab Injection; Drug: Paclitaxel injection

INTERVENTIONS:
Biological: LVGN6051 Monoclonal Antibody Injection — LVGN6051 Monoclonal Antibody Injection:1 mg/kg or 2 mg/kg, every 3 weeks(Q3W) , on the first day of the treatment cycle for up to 2 years.
  Other Names: LVGN6051
Biological: toripalimab Injection — toripalimab Injection: 240mg fixed dose,Q3W, on the first day of the treatment cycle for up to 2 years.
Drug: Paclitaxel injection — paclitaxel Injection:5ml:100 mg/m2(80 mg/m2 or 60 mg/m2 can be used if necessary),Q3W,on the first and eighth day of the treatment cycle for up to 2 years

SUMMARY:
The purpose of this study is to assess the safety and efficacy of LVGN6051 (4-1BB agonistic antibody) combined with toripalimab (anti-PD-1 antibody) and paclitaxel (anti-tubulin chemotherapy) in patients with recurrent/metastatic head and neck squamous cell carcinoma who rapidly progress from previous neoadjuvant, curative, or adjuvant platinum-containing therapy, or who are currently contraindicated for platinum-containing treatment.

DETAILED DESCRIPTION:
This is a multicenter, open-labeled, single-arm Phase 2 clinical study to evaluate the safety and efficacy of LVGN6051 in combination with toripalimab and paclitaxel in selected patients with recurrent/metastatic head and neck squamous cell carcinoma under the guidance of Good Clinical Practise(GCP).

This study comprises two parts. Part 1 (Safety run-in Phase) is designed to confirm the dose of combination therapy in Part 2. Part 1 includes a "3+3 dose-escalation design" for 2 dose levels, i.e., LVGN6051 1 mg/kg or LVGN6051 2 mg/kg with standard doses of toripalimab and paclitaxel (every 3 weeks for a treatment cycle). Part 1 will treat up to 12 DLT-evaluable patients, and the Data monitoring committee(DMC), based on the safety profile, will confirm the recommended dose for combination therapy in Part 2.

Part 2 (Efficacy Exploration Phase) will treat up to 52 patients with evaluable tumor response (efficacy) using the recommended dose of combination therapy determined in Part 1. The sample size for Part 2 is based on Simon's two-stage minimax design, which uses the Response Evaluation Criteria in Solid Tumors (RECIST 1.1) objective response rate (ORR) as the primary efficacy endpoint. The first stage will include 28 patients with evaluable tumor response (efficacy). If 6 or more responses are observed, the second stage 2 will consist of an additional 24 patients with evaluable tumor response. Part 1 patients with the same dose level as Part 2, if they meet evaluable tumor response, can be included in the required 52 patients with evaluable tumor response.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18 years or older on the date of signing the informed consent.
2. Understand and be willing to sign a written informed consent.
3. Patients with recurrent/metastatic head and neck squamous cell carcinoma confirmed by histology or cytology (the primary tumor is located in the oral cavity, oropharynx, hypopharynx, or larynx) that cannot be resected and cannot be cured by local treatment.
4. The status of head and neck squamous cell carcinoma meets one of the following requirements: a. There is still residual tumor, local recurrence, or metastatic cancer within 6 months after platinum-containing neoadjuvant treatment, adjuvant treatment, or curative concurrent chemoradiotherapy, or b. Any residual tumor, local recurrence, or metastatic cancer should receive first-line systemic therapy, but this first-line systemic therapy is not suitable for platinum-containing regimens.
5. Have measurable lesions as defined by the RECIST 1.1.
6. ECOG PS 0 or 1.
7. Life expectancy estimated at ≥3 months.
8. The functions of important organs within 1 week before the first dose meet all the following requirements: a. Hb ≥9.0 g/dL (90 g/L), b. ANC ≥1500/μL (1.5×109/L), c. Platelet count (PLT) ≥100,000/μL (100×109/L), d. Total bilirubin ≤ upper limit of normal laboratory value (ULN), e. AST ≤1.5× ULN and ALT ≤1.5× ULN, f. International normalized ratio (INR)/prothrombin time (PT) and activated partial thromboplastin time (aPTT) ≤1.5× ULN, g. Serum amylase and lipase ≤1.5× ULN, h. serum albumin ≥3.0 g/dL (30 g/L), and i. CCR ≥30 ml/min.
9. Female patients of childbearing potential should have a negative blood pregnancy test or urine pregnancy test within 72 hours before the first dose of study treatment.
10. Male patients should agree to take adequate contraceptive measures from the first dose of study treatment to 180 days after the last dose.

Exclusion Criteria:

1. Have received drug treatment targeting CD137 (4-1BB) or paclitaxel injection.
2. Subjects who are suitable to receive curative-intent local treatment.
3. Have received any systemic anti-tumor treatment after disease recurrence or metastasis.
4. Failed to fully recover from the adverse events caused by the previous anti-tumor treatment within 2 weeks before receiving the first dose of study treatment (i.e., ≤ grade 1 or baseline).
5. At the first dose of study treatment, it is still within 5 half-lives of previous anti-cancer agents.
6. Have risk of rapidly progressive disease, immediate risk of massive bleeding, airway obstruction, or uncontrolled significant tumor pain that, in the opinion of the investigator, may impair compliance with study treatment.
7. Diagnosed with immunodeficiency or receiving systemic steroids or any other immunosuppressive treatments within 7 days before the first dose of study treatment. The use of inhaled, topical, or physiologic doses of corticosteroids is allowed, i.e., ≤10 mg/day of prednisone or equivalent.
8. Have other malignant tumors diagnosed and/or treated within 5 years before the first dose of study treatment, except for cured basal cell carcinoma of the skin, cured squamous cell carcinoma of the skin, resected uterine cervical carcinoma in situ, resected breast cancer in situ. Other exceptions can be discussed with the sponsor.
9. Known occurrence of active central nervous system (CNS) metastases and/or cancerous meningitis.
10. Have an active autoimmune disease that has required systemic treatment, such as disease-modifying agents, corticosteroids, or immunosuppressive drugs in the past 2 years. Replacement therapies (such as thyroxine, insulin, or physiological corticosteroid replacement therapy for hypothyroidism, adrenal insufficiency, pituitary insufficiency, etc.) are not considered systemic treatments.
11. Have previously received allogeneic tissue/organ transplantation or any cell therapy.
12. Currently suffering from active, non-infectious pneumonia or interstitial lung disease that requires treatment with oral or intravenous glucocorticoids.
13. Active infection requiring intravenous (IV) anti-infective drugs within the first 14 days before the first dose of study treatment or the presence of unhealed wounds or ulcers.
14. The investigator believes that any previous or existing medical condition, treatment, or laboratory test abnormality may affect the study results, interfere with the patient's participation in the entire study, or the study participation is not in the patient's best interest.
15. Female patients who are pregnant or nursing or who plan to become pregnant or give birth during the study period (i.e., from the beginning of the screening period to 180 days after the last treatment).
16. Patients known to have tested positive for human immunodeficiency virus (HIV) or known to have acquired immunodeficiency syndrome (AIDS).
17. Known to have active hepatitis B or hepatitis C.
18. Have received live virus vaccine within 30 days before the first dose of study treatment.
19. Have received systemic immune-stimulating drugs (e.g., IL-2, IFN-γ) within 4 weeks before the first dose of study treatment.
20. Clinically significant heart and CNS disorders, including acute myocardial infarction within 6 months before Cycle 1 Day 1, congestive heart failure as Class III or IV by the New York Heart Association, unstable angina, uncontrolled arrhythmias requiring further treatment, stroke, or brain hemorrhage. Subjects with arrhythmia who are treated with antiarrhythmic drugs and whose electrocardiogram (ECG) screening shows a controlled heart rhythm may be enrolled.
21. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage.
22. Patients with a history of severe allergies may be allergic to the ingredients of the investigational drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-06-21 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
to determine treatment-related adverse events (TRAEs, the safety and tolerability of two preset dose levels ) | 6 months
  The safety and tolerability of two preset dose levels based on treatment-related adverse events (TRAEs), including dose-limiting toxicities(DLTs )and serious adverse events (SAEs), through a "safety run-in" to determine the Part 2 therapeutic dose of LVGN6051 in combination with toripalimab and paclitaxel. (Part 1)
to determine objective response rate (ORR) | through study completion, an average of 30 months
  The anti-tumor activity of LVGN6051 combined with toripalimab and paclitaxel will be evaluated by independent central review (ICR) according to RECIST 1.1 for objective response rate (ORR). (Part 2)

CONTACTS AND LOCATIONS:
Overall Officials: Ye Guo, Principal Investigator — Shanghai Oriental Hospital
Locations (16):
- China (16):
  - Anhui Cancer Hospital, Hefei, Anhui
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Beijing Tongren Hospital Affiliated to Capital Medical University, Beijing, Beijing Municipality
  - Fujian cancer hospital, Fuzhou, Fujian
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Guangxi Medical University Cancer Hospital, Nanning, Guangxi
  - Henan cancer hospital, Zhengzhou, Henan
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Xiangya Hospital Central South University, Changsha, Hunan
  - The Second Xiangya Hospital, Central South University, Changsha, Hunan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Liaoning cancer hospital, Shenyang, Liaoning
  - Shanghai Oriental Hospital, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang